CLINICAL TRIAL: NCT00887120
Title: Pharmacokinetics and Efficacy of Low- or Standard-dose of Lopinavir/Ritonavir (Kaletra®) in PI-naïve HIV-1 Infected Children
Brief Title: Dose Reduction of Lopinavir in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Ministry of Education, Thailand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIV-NAT045
Record Dates: First submitted 2009-04-21; First posted 2009-04-23 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: HIV Infections
Keywords: Second line treatment; therapeutic drug monitoring; Asia; LPV; children; pharmacokinetic; To study the pharmacokinetics of low-dose and standard dose, lopinavir/ritonavir in Protease inhibitor (PI)- naive HIV-1 infected Thai patients.; To study clinical and immunological efficacy after 48-weeks of lopinavir/ritonavir-based antiretroviral therapy in PI naive HIV-1 infected Thai patients.
MeSH Terms: conditions — HIV Infections | interventions — Lopinavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Lopinavir/ritonavir standard dose + zidovudine and lamivudine
  Interventions: Drug: Lopinavir/ritonavir standard dose According to WHO simplified dosing table
- 2 (Active Comparator): Lopinavir/ritonavir low dose (70% of standard dose) + zidovudine and lamivudine
  Interventions: Drug: Lopinavir/ritonavir low dose ( 70% of WHO recommended dosing table)

INTERVENTIONS:
Drug: Lopinavir/ritonavir standard dose According to WHO simplified dosing table — * BW 6-7.9 kg: 1.5 mL oral q 12 hr
  * BW 8.0-16.9 kg: 2.0 ml oral q 12 hr
  * BW 17.0-19.9 kg: 2.5 ml oral q 12 hr
  * BW 20.0 - 24.9 kg: 3.0 ml oral q 12 hr
  * BW 25.0 - 29.9 kg: 3.5 ml oral q 12 hr
  * BW 30.0-34.9 kg: 4.0 ml oral q 12 hr
  * BW > 35 kg: 5.0 ml oral q 12 hr
  Dose of Zidovudine (AZT) is 180-240 mg/m2 per dose every 12 hours Dose of Lamivudine (3TC) is 4 mg/kg every 12 hours Dose of Lopinavir/ritonavir (LPV/r)
  Arms: 1
Drug: Lopinavir/ritonavir low dose ( 70% of WHO recommended dosing table) — * BW 6-7.9 kg: 1.0 mL oral q 12 hr
  * BW 8.0-16.9 kg: 1.5 ml oral q 12 hr
  * BW 17.0-19.9 kg: 1.8 ml oral q 12 hr
  * BW 20.0 - 24.9 kg: 2.0 ml oral q 12 hr
  * BW 25.0 - 29.9 kg: 2.5 ml oral q 12 hr
  * BW 30.0-34.9 kg: 3.0 ml oral q 12 hr
  * BW > 35 kg: 3.5 ml oral q 12 h
  Dose of Zidovudine (AZT) is 180-240 mg/m2 per dose every 12 hours Dose of Lamivudine (3TC) is 4 mg/kg every 12 hours Dose of Lopinavir/ritonavir (LPV/r)
  Arms: 2

SUMMARY:
To study the pharmacokinetics of low-dose and standard dose, lopinavir/ritonavir in ARV PI naive HIV-1 infected Thai children.

To study clinical and immunological efficacy after 48 weeks of lopinavir/ritonavir in PI naïve HIV-1 infected Thai children

DETAILED DESCRIPTION:
In 2002, the Thai Ministry of Public Health (MOPH) launched the National Access to Antiretroviral Program for People living with HIV/AIDS (NAPHA) with the aim of providing treatment to all Thai patients who needed antiretroviral treatment. By the end of 2005, 80,000 HIV-infected Thais were treated in the NAPHA program, including about 6,000 children. The antiretroviral treatment regimen consists of three antiretroviral drugs (ARV). The first-line regimen used in NAPHA are mainly generic drugs produced by Thai government pharmaceutical organization (GPO), including a fixed-drug combination of stavudine, lamivudine, and nevirapine (GPOvir);and a fixed-drug combination of zidovudine, lamivudine, and nevirapine (GPOvir-Z). Majority of patients respond very well with first-line regimen(1,2), however about 15% of patients have drug resistance to first-line regimen and require second-line regimen(3). The protease inhibitors (PIs) is used as a second-line regimen, however there are limitations in terms of cost and metabolic complications(4).

Lopinavir/ritonavir is the most widely use protease inhibitors in children because of its high efficacy and a syrup formulation that easy to use in small children. There is evidence supported that the recommended dose according to US-FDA or EU guidelines resulting in much higher plasma blood level in Thai children. Data from 19 Thai children demonstrated Cmin of 5.9 mg/L compare to 3.4 mg/L in US children when use the same dose (the minimum acceptable Cmin is 1.0 mg/L) (5,6). There is a study HIVNAT019, which demonstrated acceptable LPV plasma concentration and treatment outcome in Thai HIV-infected adult when use reduced dose of LPV/r 266mg/66 mg compare to standard dose of 400mg/100mg (7).

Therefore, the study of pharmacokinetic of low dose of LPV/r in Thai HIV-infected children is very important to assess the safety and efficacy of this strategy. This will lead to appropriate ARV dose in children to reduce long-term adverse events, and also reduce the ARV cost.

ELIGIBILITY:
Inclusion Criteria:

* Age from 2- 18 years old
* Documented positive test for HIV-1 infection
* PI-naïve
* HIV RNA viral load > 1,000 copies
* Written informed consent

Exclusion Criteria:

* Active opportunistic infection
* Relevant history or current condition, illness that might interfere with drug absorption, distribution, metabolism or excretion.
* Use of concomitant medication that may interfere with the pharmacokinetics of lopinavir/ritonavir
* Pregnancy or lactating
* Inability to understand the nature and extent of the study and the procedures required.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2007-04; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
pharmacokinetics of standard vs low dose LPV/r | 4 weeks after start ART

SECONDARY OUTCOMES:
efficacy and safety of standard and low dose LPV/r | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kiat Ruxrungtham, MD, Principal Investigator — Department of Medicine, Faculty of Medicine, Chulalongkorn University and Thai Red Cross Aids Research Centre - HIV-NAT
Locations (1):
- HIV-NAT, Thai Red Cross AIDS Research Center, Bangkok, Bangkok, Thailand

REFERENCES:
- [Derived] Puthanakit T, van der Lugt J, Bunupuradah T, Ananworanich J, Gorowara M, Phasomsap C, Jupimai T, Boonrak P, Pancharoen C, Burger D, Ruxrungtham K. Pharmacokinetics and 48 week efficacy of low-dose lopinavir/ritonavir in HIV-infected children. J Antimicrob Chemother. 2009 Nov;64(5):1080-6. doi: 10.1093/jac/dkp322. Epub 2009 Sep 2. PMID 19729375
- See also: HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org